CLINICAL TRIAL: NCT05379764
Title: A Randomized Controlled Single Blind Parallel Study, Evaluating Embodiment in a VR Scenario Designed to Elicit Stress in a Return to Work E-vironment.
Brief Title: VR Embodiment for Stress Evaluation in a Return to Work Simulation
Acronym: VRSTEVAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinique Saint-Jean, Bruxelles (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Dr. Arnaud Bosteels, Medical Doctor, Clinique Saint-Jean, Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: VRSTEVAR01
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Virtual Reality; Stress; Burnout
Keywords: Virtual reality; stress; embodiment; Burnout
MeSH Terms: conditions — Burnout, Psychological | interventions — Observation

STUDY DESIGN:
Intervention Model Description: Parallel single blind randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator and outcome assessor will have no idea who is in what arm. It will be another investigator who is randomising the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embodiment group (Experimental): This group this group will view the VR scenario being 'embodied' in the avatar who is experiencing the VR scenario. This implies first persons perspective, agency over the avatar, multi-sensorial integration and co-location.
  Interventions: Other: Embodiment
- observation group (Sham Comparator): This group will view the VR scenario from a third persons perspective , as an observer.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Embodiment — Embodiment of a real human in a virtual human (avatar) means that the real human feels incarnated in the avatar. This happens when the real human sees the VRscenario from first person perspective, that the real human can make the avatar move (=agency over the avatar), multi-sensorial integration (=there is a link between the brain of the real human and the avatar. Example, when the avatar sits on a chair, the real human will too and he feels that he is sitting on a chair. Or when the avatar is moving the real human is doing the same movement (and of course the brain of the real human is aware of this movement)) and co-location (= avatar and real human have the sane posture).
  Arms: Embodiment group
Other: Observation — The person is looking at the VR scenario as if s/he was looking at a TV
  Arms: observation group

SUMMARY:
Comparing the emotional effect of two different versions of one VR experience. The VR experience will simulate a typical return to work situation after an absence due to burnout.

The difference of the VR scenario is the point of view. In the first version, the 'standard' version, the user is looking at the VR experience from a neutral point of view, as if s/he was watching a 2D screen. In the second version, the 'embodiment' version, a VR features is added to have the user feeling incarnated in a digital human. This will enhance the feeling of being present in the virtual world and will enhance the emotional answer. The measured endpoint will be the evoked emotions, in particular stress.

ELIGIBILITY:
Inclusion Criteria:

* working in the office building where the study will be conducted

Exclusion Criteria:

* neurologic disorder precluding the use of VR goggles (epilepsy, …),
* facial wounds precluding the use of VR goggles.
* a preliminary test evaluating the stress level will be conducted, DASS -21: stress levels above moderate is an exclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
measured stress level | this will be evaluated after the intervention and will take 15 min.
  This is measured with a Visual Analogue Scale from 1-10 and with the DASS-21, subscale stress

SECONDARY OUTCOMES:
measured Emotional level | 15 min, before (baseline) and after the intervention
  general emotional level, measured with the PANAS scale
measured stress baseline | 15min, before the intervention
  This is measured with a Visual Analogue Scale from 1-10 and with the DASS-21, subscale
embodiment evaluation | 20 min after the intervention
  measuring the level of embodiment experienced by the user
plausibility illusion and place illusion | 20 min after intervention
  Answering the question: is it possible that it happens and that it happens here?. Assessed together with the level of embodiment, also with a questionnaire.

IPD SHARING:
Plan to Share IPD: No